CLINICAL TRIAL: NCT04638205
Title: The Life Paths That Lead Teenagers to Attempted Suicide: Trajectories of Proximal Adversity
Brief Title: The Life Paths That Lead Teenagers to Attempted Suicide:Trajectories of Proximal Adversity
Acronym: TAPAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_20; 2018-A03065-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-07-09; First posted 2020-11-20 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Suicide, Attempted
Keywords: Suicide attempt; adolescence; adverse life event; developmental model; trajectories
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suicide attempt cases: Adolescents and young adults who attempted suicide between 7 and 30 days prior the inclusion
- Non-suicidal controls: Adolescents and young adults without history of suicide attempt or ideation

SUMMARY:
Suicidal behaviors seriously alter the vital and functional prognosis of adolescents. Although the literature has lighted out a considerable number of risk factors for suicide attempts in youth, theoretical models - among which bio-psycho-social models - still lack empirical evidence. More specifically, the way adverse life events dynamically interact together and with the individual's diathesis to precipitate suicidal attempts remains unclear. Studies of life trajectories have opened an alternative approach to traditional linear epidemiological analysis to capture such a complex process. To date, adverse trajectories approaches never have been applied to the period immediately preceding the occurrence of the suicidal gesture (proximal adverse trajectories).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for cases
* Youth aged 15-24 inclusive
* Who stayed at the hospital or in the emergency room for less than 15 days after a first suicide attempt
* Who were discharged less than 15 days ago
* Who gave their informed consent for majors, or whose parents gave their informed consent for minors Inclusion criteria for controls
* Youth aged 15-24 inclusive
* Who have never experienced any suicidal ideation or suicide attempt
* Who gave their informed consent for majors, or whose parents gave their informed consent for minors Inclusion criteria for informants
* Close relatives of the participant
* Who are major
* Who lived in the same household as the participant or have interacted with him/her for more than half the weeks of the year preceding the index suicide attempt

Exclusion Criteria:

* No consent or consent withdrawal for majors and/or their parents for minors
* Neurological or psychiatric condition altering the capacity to understand

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient recruitment will be supported by the VigilanS program. VigilanS is a suicide recurrence prevention device implemented in all establishments in the Hauts-de-France region that receive patients who have attempted suicide (www.dispositifvigilans.org).
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Growth parameters of the patterns of proximal adverse trajectories in adolescents who attempted suicide, as compared to non-suicidal adolescents | 1 year
  We will build growth mixture models to account for the 1-year longitudinal evolution of the Burden of Adversity values. Each group will be characterized by the parameters (intercepts and slopes) of the best-fitting model.
  We will the compare the parameters of the 2 groups to search for statistical differences

SECONDARY OUTCOMES:
Statistical tests comparing the sociodemographic, vulnerabily and psychopathological indicators between the sub-group of adolescents identified from the mixture model. | 1 year
  Growth mixture models will allow for identifying sub-groups of individuals who are similar as regards to their burden of adversity trajectories. We will compare the characteristics of theses subgroups
Growth parameters of the patterns of evolution of psychological pain | 1 year
  Parallel to the burden of adversity growth models, we will build, for each group, growth models to predict the longitudinal evolution of psychological pain.
  We will then test whether the growth parameters of the ideation/pain trajectories correlate with those of the adversity trajectories
Growth parameters of the patterns of evolution of suicidal ideation intensity | 1 year
  Parallel to the burden of adversity growth models, we will build, for each group, growth models to predict the longitudinal evolution of the severity of the suicidal ideations.
  We will then test whether the growth parameters of the ideation/pain trajectories correlate with those of the adversity trajectories

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Edouard Notredame, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Fontan - Chu Lille, Lille, France